CLINICAL TRIAL: NCT05786807
Title: Effect of H. Pylori Eradication on Alleviating Symptoms in Functional Dyspepsia Patients: A Multicenter, Comparative Study
Brief Title: Effect of H. Pylori Eradication on Alleviating Symptoms in Functional Dyspepsia Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Suck Chei Choi, Coordinating Investigator, Wonkwang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCAB_004
Record Dates: First submitted 2023-02-24; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Helicobacter Pylori-positive With Functional Dyspepsia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tegoprazan 50mg (Experimental): single group
  Interventions: Drug: K-CAB

INTERVENTIONS:
Drug: K-CAB — Tegoprazan 50 mg 1 tab twice daily Amoxicillin 500mg 2 cap twice daily Clarithromycin 500mg 1tab twice daily

SUMMARY:
In patients with Helicobacter pylori-positive functional dyspepsia, long-term follow-up for 6 months after standard triple therapy first-line eradication treatment, the rate of symptom disappearance and degree of improvement of functional dyspepsia were confirmed through changes in symptom scores and changes in drug usage, and eradication treatment The purpose of this study is to confirm the rate of symptom disappearance according to the results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of 19 and 75
* Who have symptoms of functional dyspepsia (early fullness, postprandial discomfort, epigastric pain, epigastric soreness) that correspond to Rome criteria 4 (diagnostic criteria questionnaire)

Exclusion Criteria:

* Small intestine and large intestine disease within 6 months of the screening visit (Visit 1)
* liver, pancreatobiliary disease within 6 months of the screening visit (Visit 1)
* peptic ulcer within 6 months of the screening visit (Visit 1)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of disappearance of dyspepsia symptoms | Day 176
  Rate of disappearance of dyspepsia symptoms after 6 months of eradication treatment

SECONDARY OUTCOMES:
Improvement rate of dyspepsia symptoms | Day 92, Day 176
  Change rate of dyspepsia symptoms after 3 months and 6 months of eradication treatment
Number of days of dyspepsia drug administration | Day 92, Day 176
  Number of days of dyspepsia drug administration after 3 months and 6 months of eradication treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suck Chei Choi, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwang University Hospital, Iksan, Jeollabuk, South Korea